CLINICAL TRIAL: NCT01479829
Title: Cyclooxygenase-2-Inhibitor Combination Treatment for Bipolar Depression: Role of Inflammation and Kynurenine Pathway Biomarkers
Brief Title: Cyclooxygenase-2-Inhibitor Combination Treatment for Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Angelos Halaris, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 203368
Record Dates: First submitted 2011-09-22; First posted 2011-11-24 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression; Celecoxib; Escitalopram; Inflammation
MeSH Terms: conditions — Bipolar Disorder; Inflammation | interventions — Escitalopram; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention cohort (Experimental): Participants assigned to the intervention cohort receive 10mg escitalopram twice daily plus 200mg celecoxib twice daily.
  Interventions: Drug: Escitalopram; Drug: Celecoxib
- Control cohort (Placebo Comparator): Participants assigned to the control cohort receive 10mg escitalopram twice daily plus placebo administered twice daily.
  Interventions: Drug: Escitalopram; Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram is a Selective Serotonin Reuptake Inhibitor (SSRI)
  Other Names: Lexapro
Drug: Celecoxib — Celecoxib is a nonsteroidal anti-inflammatory drug
  Other Names: Celebrex
  Arms: Intervention cohort
Drug: Placebo — Placebo is a manufactured capsule with no active ingredient
  Other Names: Inactive drug
  Arms: Control cohort

SUMMARY:
This project will attempt to enhance and augment the antidepressant efficacy of a commonly used antidepressant in poorly responding bipolar depressed patients.

DETAILED DESCRIPTION:
This is a placebo-controlled study of patients with bipolar I disorder (BPD) utilizing a well-known antidepressant, escitalopram (ESC), in combination with the anti-inflammatory agent, celecoxib (CBX). The investigators hypothesize that combination treatment will lead to a qualitatively and quantitatively augmented response and will result in greater numbers of remitters compared to ESC monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 - 65 years old at time of screening visit. Both genders and any race will be accepted.
* Diagnosis of BPD I or II without significant co-morbid secondary medical or psychiatric diagnoses; no substance abuse or dependence during preceding 12 months
* A minimum score of 18 on the first 17 items of the 21-item Hamilton Depression Scale
* Willingness to washout for a reasonable time (depending on the substance) from: Vitamin E and fish oils (>600 IU/day), non-aspirin NSAIDs or aspirin (>81 mg/day, H2 receptor antagonists, Ginko biloba, caffeine on morning of blood drawing, and to institute lights-out at 23:00 hours on the nights before blood drawings

Exclusion Criteria:

* Any abnormal findings on the physical exam, ECG, blood/urine or minor infections
* Any pre-existing physical pain condition, including fibromyalgia
* History of peptic ulcer complicated by perforation, hemorrhage, or obstruction; symptoms of peptic ulcer within 4 weeks of enrollment date
* Any substance abuse or dependence during the preceding 12 months
* Clinically significant hypertension, anemia, liver disease, kidney disease, arthritis, diabetes, recurrent migraines, epilepsy, stroke, gum disease, autoimmune disease
* Current use of lithium
* Current use of a stimulant
* Certain steroids including use of hormonal birth control and any systemic or topical corticosteroids (hormone replacement therapy will be allowed)
* Unwillingness to refrain from H2 receptor antagonists, non-aspirin NSAIDs, or aspirin (more than 1 mg/day).
* Use of any anticoagulant agents
* Use of nicotine-containing substances. Subjects who quit smoking more than 3 months prior to assessment may be considered for the study
* Known sensitivity or allergy to the study medications or a need to receive agents that are contra-indicated in combination with CBX or ESC
* Unwillingness to fast and abstain from caffeine on mornings of blood drawings
* A sleep disorder other than insomnia or hypersomnia as a distinct symptom of major depressive disorder (MDD)
* Inability to commit to the follow-up visits between 8 and 11 am

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03-23 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Halaris, MD, PhD, Principal Investigator — Loyola Univeristy Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murata S, Murphy M, Hoppensteadt D, Fareed J, Welborn A, Halaris A. Effects of adjunctive inflammatory modulation on IL-1beta in treatment resistant bipolar depression. Brain Behav Immun. 2020 Jul;87:369-376. doi: 10.1016/j.bbi.2020.01.004. Epub 2020 Jan 7. PMID 31923551
- [Derived] Halaris A, Cantos A, Johnson K, Hakimi M, Sinacore J. Modulation of the inflammatory response benefits treatment-resistant bipolar depression: A randomized clinical trial. J Affect Disord. 2020 Jan 15;261:145-152. doi: 10.1016/j.jad.2019.10.021. Epub 2019 Oct 13. PMID 31630035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an outpatient psychiatric clinic
Pre-assignment Details: One-hundred subjects consented to participate in this study. Among these individuals, 27 participants were screen failures and eight participants withdrew prior to randomization. The remaining 65 participants were randomized and took at least one study capsule
Period: Overall Study
Arm/Group | Intervention Cohort | Control Cohort
Started | 35 | 30
Completed | 27 | 20
Not Completed | 8 | 10
Not completed — Withdrawal by Subject | 8 | 10

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all patients who were randomized and completed at least eight consecutive weeks of assigned treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Cohort | Control Cohort | Total
Number analyzed (Participants) | 27 | 20 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.48 (10.73) | 46.15 (13.50) | 42.32 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 12 | 7 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-described race: White | 19 | 13 | 32
  Self-described race: non-White | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 27 | 20 | 47

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment
Description: Participants complete the Hamilton Depression Rating Scale (HDRS-17). The HDRS-17 is a clinician-administered assessment scale measuring the melancholic and physical symptoms of depression. Possible scores range from 0 to 54 (i.e., where higher scores indicate worse depression). In this study, response to treatment is defined as a reduction in the HDRS-17 score of at least 50% after 8 weeks of treatment.
Time Frame: 8 weeks
Population: The analysis population is defined as all participants who completed at least eight weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cohort | Control Cohort
Number analyzed (Participants) | 27 | 20
Participants
  Response | 21 | 9
  No Response | 6 | 11
Statistical Analysis 1: Comparison: Intervention Cohort vs Control Cohort; The null hypothesis is that there is no difference in the response rate between patients assigned to the intervention cohort or control cohort; Test type: Superiority; p = .02, Chi-squared; Chi-square value = 5.3466 — The chi-square value with 1 degree of freedom was 5.3466

2. Primary Outcome: Disease Remission
Description: Participants complete the Hamilton Depression Rating Scale (HDRS-17). The HDRS-17 is a clinician-administered assessment scale measuring the melancholic and physical symptoms of depression. Possible scores range from 0 to 54 (i.e., where higher scores indicate worse depression). In this study, diisease remission is defined as an HDRS-17 score less than 8 points after 8 weeks of treatment.
Time Frame: 8 weeks
Population: The analysis population is defined as all participants who completed at least eight weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cohort | Control Cohort
Number analyzed (Participants) | 27 | 20
Participants
  Remission | 17 | 2
  No Remission | 10 | 18
Statistical Analysis 1: Comparison: Intervention Cohort vs Control Cohort; The null hypothesis is that there is no difference in the remission rate between patients assigned to the intervention cohort or control cohort; Test type: Superiority; p < .001, Chi-squared; Chi-square value = 13.3821 — The chi-square value with 1 degree of freedom was 13.3821

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention Cohort | Control Cohort
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/30
Other Adverse Events (participants affected / at risk) | 0/35 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-01-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT01479829/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT01479829/ICF_001.pdf